CLINICAL TRIAL: NCT00279500
Title: Chronic Retinal Electrodes to Provide Electrical Stimulation of the Retina to Elicit Visual Percepts in Blind Subjects
Brief Title: Feasibility Study of a Chronic Retinal Stimulator in Retinitis Pigmentosa
Acronym: (A16)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0002
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2018-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Subjects with a confirmed history of advanced retinal degenerative disease and meeting the inclusion criteria listed will be considered as eligible participants in the study. Subjects who have a condition listed in the exclusion criteria will not be allowed to participate in the study. Eligible subjects with the above diagnoses will be recruited from the Doheny Eye Institute at the University of Southern California. Additionally, new subjects encountered in the clinic who fulfill the inclusion criteria will also be eligible to participate. Upon meeting the entry criteria, all subjects must sign an Informed Consent prior to enrollment in the study. Since the subjects are blind, an individual not associated with this study must read the informed consent to the subject. This person must sign the consent form as a witness to the informed consent process.
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Experimental): Argus 16 Retinal Stimulation System-single arm study.
  Interventions: Device: Argus 16 Retinal Stimulation System

INTERVENTIONS:
Device: Argus 16 Retinal Stimulation System — The chronic retinal stimulation system is an implantable electronic device designed to provide electrical stimulation of the retina in order to elicit visual percepts in blind subjects.

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the retinal stimulation system by evaluating the data after chronic implantation.

DETAILED DESCRIPTION:
The chronic retinal stimulation system is an implantable electronic device designed to provide electrical stimulation of the retina in order to elicit visual percepts in blind subjects.

This chronic feasibility study will evaluate the ability of subjects to resolve multiple percepts and patterns under various stimulus conditions and optimize the effectiveness of electrical stimulus parameters with an initial chronic design.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed history of retinal degenerative disease in the worse seeing eye with remaining vision no better than light perception. The fellow eye can have any visual acuity but must have better vision than the eye that will have the surgery.
* History of former useful form vision in worse-seeing eye
* Acceptable ability to describe visual percepts
* Age eighteen (18) or older

Exclusion Criteria:

* History of glaucoma
* Optic neuropathy or other confirmed damage to optic nerve or visual cortical damage
* Presence of communicable disease/infection
* Pregnancy
* History of claustrophobia
* Inconsistent flash detection thresholds
* Any other diseases that can effect the function of the retina
* Subjects with a Beck Depression Inventory Interpretation score of >30 and subsequent diagnosis of depression by a psychiatrist.
* Corneal degeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2002-02-27 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Olmos, MD, Principal Investigator — Doheny Eye Institute
Locations (1):
- Doheny Eye Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yue L, Wuyyuru V, Gonzalez-Calle A, Dorn JD, Humayun MS. Retina-electrode interface properties and vision restoration by two generations of retinal prostheses in one patient-one in each eye. J Neural Eng. 2020 Apr 9;17(2):026020. doi: 10.1088/1741-2552/ab7c8f. PMID 32131056
- [Derived] Nanduri D, Fine I, Horsager A, Boynton GM, Humayun MS, Greenberg RJ, Weiland JD. Frequency and amplitude modulation have different effects on the percepts elicited by retinal stimulation. Invest Ophthalmol Vis Sci. 2012 Jan 20;53(1):205-14. doi: 10.1167/iovs.11-8401. PMID 22110084
- [Derived] Eng JG, Agrawal RN, Tozer KR, Ross-Cisneros FN, Dagnelie G, Greenberg RJ, Chader GJ, Weiland JD, Rao NA, Sadun AA, Humayun MS. Morphometric analysis of optic nerves and retina from an end-stage retinitis pigmentosa patient with an implanted active epiretinal array. Invest Ophthalmol Vis Sci. 2011 Jun 28;52(7):4610-6. doi: 10.1167/iovs.09-4936. PMID 21296811
- [Derived] Horsager A, Boynton GM, Greenberg RJ, Fine I. Temporal interactions during paired-electrode stimulation in two retinal prosthesis subjects. Invest Ophthalmol Vis Sci. 2011 Feb 1;52(1):549-57. doi: 10.1167/iovs.10-5282. Print 2011 Jan. PMID 20720224
- [Derived] Greenwald SH, Horsager A, Humayun MS, Greenberg RJ, McMahon MJ, Fine I. Brightness as a function of current amplitude in human retinal electrical stimulation. Invest Ophthalmol Vis Sci. 2009 Nov;50(11):5017-25. doi: 10.1167/iovs.08-2897. Epub 2009 Jul 15. PMID 19608533
- [Derived] Caspi A, Dorn JD, McClure KH, Humayun MS, Greenberg RJ, McMahon MJ. Feasibility study of a retinal prosthesis: spatial vision with a 16-electrode implant. Arch Ophthalmol. 2009 Apr;127(4):398-401. doi: 10.1001/archophthalmol.2009.20. PMID 19365014
- [Derived] Horsager A, Greenwald SH, Weiland JD, Humayun MS, Greenberg RJ, McMahon MJ, Boynton GM, Fine I. Predicting visual sensitivity in retinal prosthesis patients. Invest Ophthalmol Vis Sci. 2009 Apr;50(4):1483-91. doi: 10.1167/iovs.08-2595. Epub 2008 Dec 20. PMID 19098313
- [Derived] de Balthasar C, Patel S, Roy A, Freda R, Greenwald S, Horsager A, Mahadevappa M, Yanai D, McMahon MJ, Humayun MS, Greenberg RJ, Weiland JD, Fine I. Factors affecting perceptual thresholds in epiretinal prostheses. Invest Ophthalmol Vis Sci. 2008 Jun;49(6):2303-14. doi: 10.1167/iovs.07-0696. PMID 18515576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2002. The last subject of 6 was enrolled in June 2004.
Groups:
- Argus 16 Retinal Stimulation System: Single arm study in which all patients were implanted with the Argus 16 Retinal Stimulation System, which stimulates retinal (eye) cells.
Period: Overall Study
Arm/Group | Argus 16 Retinal Stimulation System
Started | 6 (6 patients treated)
Completed | 6 (6 patients treated)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Single arm study in which all patients were implanted with the Argus 16 Retinal Stimulation System, which stimulates retinal (eye) cells.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Visual Acuity [Count of Participants; unit: Participants]
  No Light Perception | 2
  Bare Light Perception | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events From 2 Weeks Post-op Until the End of the Study
Description: All adverse events are collected as a result of chronic electrical stimulation and/or surgical complications.
Time Frame: From 2 weeks post-op until end of device usage, up to 10 years.
Measure: Number; unit: total number of AEs
Arm/Group | Argus 16 Retinal Stimulation System
Number analyzed (Participants) | 6
total number of AEs | 34

ADVERSE EVENTS:
Time Frame: 10 years
Groups:
- Argus 16 Retinal Stimulation System: Single arm study in which all patients receive a device to stimulate retinal (eye) cells. The treatment is intended to evaluate the safety and efficacy of the retinal stimulation system by evaluating the data after chronic implantation.
Arm/Group | Argus 16 Retinal Stimulation System
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argus 16 Retinal Stimulation System (N=6)
Retinal Detachment (Eye disorders) | 2 (2)
Endophthalmitis (Eye disorders) | 1 (3)
Conjunctival Erosion (Eye disorders) | 2 (5)
Dizziness (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Mesenteric Ischemia (Gastrointestinal disorders) | 1 (1)
Re-Tack (Eye disorders) | 1 (1) — as a result of bump to the head
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argus 16 Retinal Stimulation System (N=6)
Array Rotation (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Corneal Dryness (Eye disorders) | 2 (2)
Corneal Opacity (Eye disorders) | 1 (1)
Epiretinal Membrane (Eye disorders) | 1 (2)
Headache (Eye disorders) | 1 (2)
Headache and Nausea (Eye disorders) | 1 (1)
Inflammation (Eye disorders) | 1 (1)
Numbness (Eye disorders) | 1 (1)
Ocular Pain (Eye disorders) | 1 (2)
Pain and Nausea (Eye disorders) | 1 (1)
Bump (General disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Dizziness (Eye disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Fall (with array movement) (Injury, poisoning and procedural complications) | 1 (1)
Headache (General disorders) | 3 (3)
Inflammation (General disorders) | 1 (1)
Minor Injury (right cheekbone) (Injury, poisoning and procedural complications) | 1 (1)
Mild Trauma To Head (Injury, poisoning and procedural complications) | 1 (1)
Sprained Right Wrist (Injury, poisoning and procedural complications) | 1 (1) — Motor vehicle accident
Ocular Pain (Eye disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Rash (Fluorescein Dye Reaction) (Injury, poisoning and procedural complications) | 1 (1)
Transient Ischemic Attack (Vascular disorders) | 1 (1)
Vertigo (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Separate IP agreement.